CLINICAL TRIAL: NCT00916747
Title: An Open Label Phase II Trial of Zoledronic Acid, Pravastatin, and Lonafarnib for Patients With Hutchinson-Gilford Progeria Syndrome(HGPS) and Progeroid Laminopathies
Brief Title: Study of Zoledronic Acid, Pravastatin, and Lonafarnib for Patients With Progeria
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Schering-Plough (Industry); Merck Sharp & Dohme LLC (Industry); Eiger BioPharmaceuticals (Industry)
Responsible Party: Principal Investigator, Monica E. Kleinman, Principal Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Progeria Efficacy
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Progeria
Keywords: Progeria
MeSH Terms: conditions — Progeria | interventions — lonafarnib; Zoledronic Acid; Pravastatin

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): All patients will receive zoledronic acid, pravastatin and lonafarnib
  Interventions: Drug: Lonafarnib, Zoledronic Acid, and Pravastatin

INTERVENTIONS:
Drug: Lonafarnib, Zoledronic Acid, and Pravastatin — Lonafarnib: Lonafarnib dosing will begin at 150 mg/m2 by mouth twice daily. Lonafarnib will be orally administered without planned breaks, approximately every 12 hours, for a period of 24 months. For patients unable to swallow capsules, the capsules can be opened and dissolved into Ora Blend SF or Ora-Plus.
  Zoledronic Acid: Zoledronic acid will be administered intravenously at week one, and months 6, 12, 18 and 24 of this treatment trial. Treatment will consist of one infusion over a 30 minute period.
  Pravastatin: Pravastatin will be orally administered once daily without planned breaks, approximately every 24 hours, for a period of 24 months. The drug may be taken with meals. For patients unable to swallow pills, pills can be crushed into food. Pravastatin will be dosed according to the patient weight. Patients less than 10 kg will receive 5 mg pravastatin orally, once daily. Patients weighing 10 kg or greater will receive 10 mg pravastatin daily.

SUMMARY:
Hutchinson-Gilford Progeria Syndrome (Progeria) is a rare autosomal disease that results in premature death at a median age of 13 years due to cardiovascular and cerebralvascular compromise. The mutation for this disease has been identified and results in a mutant form of lamin A that cannot be de-farnesylated. This study evaluates the combination of pravastain (a statin), lonafarnib (a farnesyltransferase inhibitor) and zoledronic acid (a bisphosphonate) in an open label phase II efficacy trial in children with Progeria. These agents all target farnesylation pathways at different points. Patients with genetically confirmed progeria will be eligible for this protocol. Treatment will be initiated for 24 months duration. Clinical and biologic parameters will be examined to assess response.

ELIGIBILITY:
Inclusion Criteria:

* Genetic Diagnosis: All patients must have confirmatory mutational analysis showing mutation in the lamin A gene.
* Clinical Diagnosis: Patients must display clinical signs of progeria as per the clinical trial team.
* Travel: Patients must be willing and able to come to Boston for appropriate studies and examinations at initiation of study and at months 6, 12, 18 and 24 on study.
* Patient must have adequate organ and marrow function as defined by the following parameters:
* Blood: APC (ANC + bands + monocytes = APC) > 1,000/microliters, Platelets > 75,000/microliters (transfusion independent); Hemoglobin >9g/dl.
* Renal: creatinine Less than or equal 1.5 times normal for age or GFR > 70 ml/min/1.73m2.
* Hepatic: bilirubin Less than or equal to 1.5 x upper limit of normal for age; SGPT (ALT) < and SGOT (AST) < 5 x normal range for age.
* PT/PTT: PT/PTT < 120% upper limit of normal OR PI approval
* No overt renal, hepatic, pulmonary disease or immune dysfunction.
* 25-hydroxyvitamin D ≥ 20 ng/ml within 4 weeks of bisphosphonate infusion.
* Signed informed consent according to institutional guidelines must be obtained and patient must begin therapy within twenty eight (28) days.

Exclusion Criteria:

* Other than the drugs used in this protocol, drugs targeted to treat Progeria are excluded. Drugs to treat symptoms of Progeria are permitted.
* Patients must not be taking medications that significantly affect the metabolism of lonafarnib at the time they start lonafarnib
* Patient must have no uncontrolled infection.
* Subjects who have known or suspected hypersensitivity to any of the excipients included in the formulation should not be treated.
* Patients must not be pregnant or breast-feeding. Female patients of childbearing potential must have negative serum or urine pregnancy test. Male and female patients of reproductive potential must agree to use a medically accepted form of birth control while on study and up to 10 weeks after treatment. It is permissible for female patients to take oral contraceptives or other hormonal methods while receiving treatment with lonafarnib.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-08; Primary Completion 2022-02 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the therapeutic effects of the combination of zoledronic acid, pravastatin and lonafarnib in patients with HGPS. | 2 years

SECONDARY OUTCOMES:
To describe any acute and chronic toxicities associated with treating progeria patients with the combination of zoledronic acid, pravastatin and lonafarnib. | 2 years
To investigate which clinical and laboratory studies are needed to monitor or alter therapy to prevent unacceptable toxicity. | 2 years
To assess the pharmacokinetics of lonafarnib in patients with progeria. | 2 years
To assay for the inhibition of HDJ-2 farnesylation in Peripheral Blood Leukocytes (PBL). | 2 years
To assay for changes in research-based potential markers of efficacy such as levels of prelamin A, mature lamin A, progerin, and HP1 in protein isolated from PBL. | 2 years
To assess changes in leptin levels, glucose utilization, skeletal abnormalities including bone mineral density and X-ray finding, joint contracture and function, and growth | 2 years
To assess changes in auditory function, dental anomalies, dermatologic changes including hair density, nutrition with calorie analysis and energy expenditure, body composition analysis by DXA scan, and cardiovascular structure and function. | 2 years
To compare and incorporate clinical and laboratory data obtain from this study with that obtained during the single agent lonafarnib trial as well as the pilot combination trial of zoledronic acid, pravastatin and lonafarnib | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kieran, MD, PhD, Principal Investigator — Children's Hospital Boston/ Dana-Farber Cancer Instittue
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Gordon LB, Norris W, Hamren S, Goodson R, LeClair J, Massaro J, Lyass A, D'Agostino RB Sr, Tuminelli K, Kieran MW, Kleinman ME. Plasma Progerin in Patients With Hutchinson-Gilford Progeria Syndrome: Immunoassay Development and Clinical Evaluation. Circulation. 2023 Jun 6;147(23):1734-1744. doi: 10.1161/CIRCULATIONAHA.122.060002. Epub 2023 Mar 15. PMID 36919608
- [Derived] Suzuki M, Jeng LJB, Chefo S, Wang Y, Price D, Li X, Wang J, Li RJ, Ma L, Yang Y, Zhang X, Zheng N, Zhang K, Joseph DB, Shroff H, Doan J, Pacanowski M, Smpokou P, Donohue K, Joffe HV. FDA approval summary for lonafarnib (Zokinvy) for the treatment of Hutchinson-Gilford progeria syndrome and processing-deficient progeroid laminopathies. Genet Med. 2023 Feb;25(2):100335. doi: 10.1016/j.gim.2022.11.003. Epub 2022 Dec 12. PMID 36507973
- [Derived] Gordon LB, Kleinman ME, Massaro J, D'Agostino RB Sr, Shappell H, Gerhard-Herman M, Smoot LB, Gordon CM, Cleveland RH, Nazarian A, Snyder BD, Ullrich NJ, Silvera VM, Liang MG, Quinn N, Miller DT, Huh SY, Dowton AA, Littlefield K, Greer MM, Kieran MW. Clinical Trial of the Protein Farnesylation Inhibitors Lonafarnib, Pravastatin, and Zoledronic Acid in Children With Hutchinson-Gilford Progeria Syndrome. Circulation. 2016 Jul 12;134(2):114-25. doi: 10.1161/CIRCULATIONAHA.116.022188. PMID 27400896
- [Derived] Gordon LB, Massaro J, D'Agostino RB Sr, Campbell SE, Brazier J, Brown WT, Kleinman ME, Kieran MW; Progeria Clinical Trials Collaborative. Impact of farnesylation inhibitors on survival in Hutchinson-Gilford progeria syndrome. Circulation. 2014 Jul 1;130(1):27-34. doi: 10.1161/CIRCULATIONAHA.113.008285. Epub 2014 May 2. PMID 24795390
- See also: The Progeria Research Foundation — http://www.progeriaresearch.org/